CLINICAL TRIAL: NCT03457025
Title: Effect of Adjuvant Hyperbaric Oxygen Therapy on Bells Palsy Outcome
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-01740
Record Dates: First submitted 2018-01-31; First posted 2018-03-07 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Bell Palsy
Keywords: Oxygen Therapy; Bells Palsy
MeSH Terms: conditions — Bell Palsy | interventions — Adrenal Cortex Hormones; Antiviral Agents; Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard of Care Therapy (Active Comparator): Reference Therapy
  Interventions: Drug: Oral Corticosteroids; Drug: Oral antivirals
- Standard of Care + HOTB (Experimental): Reference therapy in addition to Hyperbaric Oxygen Therapy
  Interventions: Drug: Oral Corticosteroids; Drug: Oral antivirals; Device: Hyperbaric Oxygen Therapy

INTERVENTIONS:
Drug: Oral Corticosteroids — Prednisone 10 day taper: 60mg for 5 days, then taper for five days to 0mg
Drug: Oral antivirals — acyclovir 400mg: one pill 4 times daily for 7 days
Device: Hyperbaric Oxygen Therapy — 2.4atm administered for twice daily dives for 5 days, 10 dives total. To be begun in the first 1 week after onset of paralysis.
  Arms: Standard of Care + HOTB

SUMMARY:
This is a randomized, single blinded, non-placebo controlled that will compare one group of Bells Palsy patients receiving the current standard of care including oral corticosteroids and oral antivirals against an experimental group receiving the current standard of care in addition to hyperbaric oxygen therapy. Outcome assessment will be based on both objective analyses of facial movements as well as subjective quality of life scales.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older exhibiting unilateral facial paralysis progressing to completion in 4 days or less.

Exclusion Criteria:

* No patients from vulnerable populations as listed above will be included.
* Subjects must be able to travel to NYULMC continually during the first 12 months following enrollment.
* During the initial visit candidates must have no associated clinical signs or symptoms consistent with other causes of facial palsy. This includes but is not limited to: auricular papules, skin rashes, parotid masses, craniofacial trauma, and the presence of other cranial or distal neuropathies excluding facial numbness, change in taste, and/or hyperacusis.
* Patients with atypical presentations will be referred for cross-sectional imaging and excluded.
* Patients with histories consistent with possible recent tick exposure, rashes, headaches, or excessive fatigue will be serologically tested for Lyme disease and excluded if it returns positive.
* Pneumothorax within the last two years is the only absolute medical exclusion criteria (FF).
* Patients who are epileptics, or are claustrophobic, will be carefully counseled on the risks of HBOT before being allowed to enroll.
* Patients with severe comorbidities will undergo evaluation by their primary care doctor and require physician approval prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Change in the percentage of subjects that return to baseline facial function 1 year following the onset of paralysis Standard of Care Group | 3, 6 and 12 months
Change in the percentage of subjects that return to baseline facial function 1 year following the onset of paralysis Standard of Care + Hyperbaric Oxygen Therapy on Bells Palsy (HBOT) Group | 3, 6 and 12 months

SECONDARY OUTCOMES:
Short Form 36 (SF-36) Score Standard of Care Group | 3, 6 and 12 months
  As part of the Medical Outcomes Study (MOS), a multi-year, multi-site study to explain variations in patient outcomes, RAND developed the 36-Item Short Form Health Survey (SF-36). The eight sections are: vitality physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health
Short Form 36 (SF-36) Score Standard of Care + HBOT | 3, 6 and 12 months
  As part of the Medical Outcomes Study (MOS), a multi-year, multi-site study to explain variations in patient outcomes, RAND developed the 36-Item Short Form Health Survey (SF-36). The eight sections are: vitality physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health
Facial Clinimetric Evaluation Scale (FaCE) Score Standard of Care Group | 3, 6 and 12 months
  Used to assess facial impairment and disability after facial paralysis. It involves 15 statements, each using a five-item Likert scale. A participant circles the most appropriate response to a given statement, whereby 1 corresponds to the lowest function and 5 corresponds to the highest function. Statements are grouped into six independent domains: social function, facial movement, facial comfort, oral function, eye comfort, and lacrimal control. A score from 0 (worst) to 100 (best) is calculated.
Facial Clinimetric Evaluation Scale (FaCE) Score Standard of Care + HBOT | 3, 6 and 12 months
  Used to assess facial impairment and disability after facial paralysis. It involves 15 statements, each using a five-item Likert scale. A participant circles the most appropriate response to a given statement, whereby 1 corresponds to the lowest function and 5 corresponds to the highest function. Statements are grouped into six independent domains: social function, facial movement, facial comfort, oral function, eye comfort, and lacrimal control. A score from 0 (worst) to 100 (best) is calculated.
Facial Disability Index (FDI) Score Standard of Care Group | 3, 6 and 12 months
  Assesses facial neuromuscular dysfunction. Consists of 10 questions regarding physical function scoring difficulty on a scale of 2-5; 5 being "no difficulty" and 2 being "much difficulty"
Facial Disability Index (FDI) Score Standard of Care + HBOT | 3, 6 and 12 months
  Assesses facial neuromuscular dysfunction. Consists of 10 questions regarding physical function scoring difficulty on a scale of 2-5; 5 being "no difficulty" and 2 being "much difficulty"

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Markey, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices). Only as pertains to study results, will be shared only during publication.
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Only shared with publication.